CLINICAL TRIAL: NCT00848107
Title: Digital Ischemic Lesions in Scleroderma Treated With Oral Treprostinil Diethanolamine: An Open-label Multicenter Extension Study
Brief Title: Open-Label Study of Oral Treprostinil in Digital Ulcers
Acronym: DISTOL-EXT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The TDE-DU-202 extension study was discontinued after the randomized, placebo-controlled TDE-DU-201 study did not meet its primary efficacy objective.
Sponsor: United Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TDE-DU-202
Record Dates: First submitted 2009-02-16; First posted 2009-02-20 (Estimated); Results first posted 2014-02-07 (Estimated); Last update posted 2024-06-18 (Actual); Status verified 2014-01

CONDITIONS: Systemic Sclerosis
Keywords: systemic sclerosis; scleroderma; digital ulcers; vasculopathy
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; digital ulcers; Vascular Diseases | interventions — treprostinil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treprostinil (Experimental): Treprostinil diethanolamine sustained release tablet initiated at 0.25 mg and titrated up to a maximum dose of 16 mg BID or the individual's maximum tolerated dose (MTD).
  Interventions: Drug: treprostinil diethanolamine

INTERVENTIONS:
Drug: treprostinil diethanolamine — sustained release tablet; BID dosing; up to 16 mg BID

SUMMARY:
This open label extension trial will allow ongoing treatment of subjects who participated in the randomized controlled trials, and will provide long term information about the safety of treprostinil diethanolamine SR in subjects with SSc and digital ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Eligible subjects who completed assessments for the final visit of the previous TDE-DU-201 controlled trial and who signed appropriate informed consent were eligible to enroll in this extension study.
* If a female of childbearing potential, the subject must have agreed to continue practicing an acceptable method of birth control (i.e., surgical sterilization, approved hormonal contraceptives, barrier methods [such as a condom or diaphragm] used with a spermicide, or an intrauterine device).

Exclusion Criteria:

* Have had any change in clinical status that, in the opinion of the Investigator, would pose a safety risk for participation in this extension study;
* Have been found to be unable to complete study assessments in the previous controlled trial;
* Have prematurely discontinued study drug during the previous study due to clinical worsening or treatment related adverse events.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 115 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Seibold, MD, Principal Investigator — Scleroderma Research Consultants LLC
Locations (26):
- United States (22):
  - University of Alabama - Birmingham - Arthritis Clinical Intervention Program, Birmingham, Alabama
  - Mayo Clinic Scottsdale, Scottsdale, Arizona
  - UCLA, Los Angeles, California
  - Barbara Davis Centre, Aurora, Colorado
  - University of Connecticut Health Center, Farmington, Connecticut
  - Georgetown University - Dept. of Medicine/Rheumatology, Washington D.C., District of Columbia
  - Northwestern University - Feinberg School of Medicine, Chicago, Illinois
  - Johns Hopkins University - Division of Rheumatology, Baltimore, Maryland
  - Boston University School of Medicine, Boston, Massachusetts
  - University of Michigan - Scleroderma Program, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - UMDNJ Clinical Research Center, New Brunswick, New Jersey
  - North Shore - LIJ Health System, Lake Success, New York
  - The Hospital for Special Surgery, New York, New York
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Toledo, Toledo, Ohio
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas - Houston, Houston, Texas
  - University of Utah, Salt Lake City, Utah
  - Virginia Mason Medical, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Canada (2):
  - St Joseph's Health Care, London, Ontario
  - Jewish General Hospital, Montreal, Quebec
- United Kingdom (2):
  - Royal Free Hospital - Center for Rheumatology, London
  - Salford Royal Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited to enroll in 26 centers in the US, Canada, and the UK in this open-label trial within 14 days of completion of TDE-DU-201. Subjects who prematurely terminated the previous controlled trial were not eligible. Data from the final study visit of the previous trial served as Baseline data and subject blinding was maintained.
Pre-assignment Details: Eligible subjects who completed assessments for the final visit of the previous controlled trial, TDE-DU-201, were eligible to enroll in this extension study. Data from this final study visit served as Baseline data. A total of 115 subjects were enrolled, with 115 subjects receiving study medication at an initial dose of 0.25 mg twice daily (BID).
Groups:
- Oral Treprostinil Diethanolamine: Oral Treprostinil Diethanolamine initiated at 0.25 mg and titrated up to a maximum dose of 16 mg BID or the individual's maximum tolerated dose (MTD).
Period: Overall Study
Arm/Group | Oral Treprostinil Diethanolamine
Started | 115
Completed | 94
Not Completed | 21
Not completed — Lost to Follow-up | 2
Not completed — Withdrawal by Subject | 8
Not completed — Adverse Event | 9
Not completed — Death | 1
Not completed — Pregnancy | 1

BASELINE CHARACTERISTICS:
Population: Efficacy was assessed using data obtained at each visit, if available, from all subjects enrolled in this study. Assessments performed after discontinuation of study drug were excluded from the summaries. All subjects who had at least one dose of study drug documented were included in the safety analysis population.
Arm/Group | Oral Treprostinil Diethanolamine
Number analyzed (Participants) | 115
Age, Continuous [Mean (Full Range); unit: years] | 50 [21 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 88
  Male | 27
Race/Ethnicity, Customized [Number; unit: participants] — *Note a subject can be included in more than one race category
  participants
    Asian | 4
    Caucasian | 97
    African-American | 13
    Native American | 1
    Not provided | 1
Years since scleroderma diagnosis [Mean (Full Range); unit: years] | 10.9 [0 to 35]
Scleroderma Classification [Number; unit: participants] — Systemic sclerosis (SSc) is commonly categorized into diffuse and limited forms but can also include the overlap syndrome (associated with other connective tissue diseases). The main distinguishing feature of the diffuse form is skin involvement proximal to the elbows and ankles and a higher risk of internal organ involvement. In limited SSc, skin involvement is confined to face, hands, feet, or forearms; however, a significant proportion of patients develop pulmonary hypertension.
  participants
    Limited | 82
    Diffuse | 33

OUTCOME MEASURES:

1. Secondary Outcome: Patient Function and QOL Measure: Scleroderma Health Assessments Questionnaire (SHAQ)- Mean Change From Study Entry in SHAQ Component Scores at Each Scheduled Assessment
Description: The SHAQ consists of 20 health assessment questionnaire questions with integer responses of 0 (without any difficulty) to 3 (unable to do), and five scleroderma-specific visual analog scale (VAS) domains (Overall Disease Activity, Raynaud's Phenomenon, Finger Ulcers, Breathing, and Intestinal Problems) with values ranging from 0.0 to 15.0 centimeters. The questions are divided into eight component domains: Dressing & Grooming, Arising, Eating, Walking, Hygiene, Reach, Grip, and Activities. Each domain score is calculated by summing the domain responses and dividing by the number of questions in that domain. Each VAS domain score is calculated by dividing the value in centimeters by 5. SHAQ component and VAS domain score ranges from 0 (least limitation) to 3 (most limitation). The aggregate SHAQ score is calculated by dividing the sum of all domain scores by 13, with a score ranging from 0 (least limitation) to 3 (most limitation).
Time Frame: Baseline and Months 1, 3, 6, and 12
Population: Efficacy was assessed by the change in net ulcer burden and in the total ulcer number from Baseline at each of the follow-up visits and the percentage of subjects with formation of new ulcers during the study. Assessments performed after discontinuation of study drug were excluded from the summaries.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Treprostinil Diethanolamine
Number analyzed (Participants) | 109
units on a scale
  Month 1 | -0.01 (0.21)
  Month 3 | 0.02 (0.23)
  Month 6 | 0.02 (0.28)
  Month 12 | -0.04 (0.27)

2. Primary Outcome: Net Ulcer Burden- Mean Change From Time of Study Entry for Each Scheduled Visit Assessment
Description: Net ulcer burden at any given assessment was defined as the number of "new" or "active" ulcers at that assessment, plus the number of "indeterminate" ulcers at that assessment that had previously been classified as either "active" or "new" at any earlier assessment during the study. The mean change in net ulcer burden from time of study entry was summarized for each scheduled visit assessment.
Time Frame: Baseline and Months 1, 3, 6, 9, 12, and 18
Population: Efficacy was assessed using data obtained at each visit, if available, from all subjects enrolled in this study. Assessments performed after discontinuation of study drug were excluded from the summaries.
Measure: Mean (Standard Deviation); unit: ulcers
Arm/Group | Oral Treprostinil Diethanolamine
Number analyzed (Participants) | 111
ulcers
  Month 1 | -0.77 (1.61)
  Month 3 | -0.52 (2.02)
  Month 6 | -0.32 (1.19)
  Month 9 | -0.52 (1.53)
  Month 12 | -0.64 (1.20)
  Month 18 | -1.67 (0.58)

3. Secondary Outcome: Patient Function and Quality of Life Measure: Cochin Hand Function Scale (CHFS)-Mean Change From Study Entry in CHFS Score at Each Scheduled Assessment
Description: The CHFS score is derived from 18 validated questions that assess functional disability and handicap due to hand involvement in rheumatoid arthritis. Each answer is scored on a scale with possible integer responses of 0(without difficulty) to 5 (impossible). The CHFS score is simply the sum of all 18 questions, divided by the number of questions actually answered, multiplied by 18. At least 10 of the 18 questions must have been answered in order for CHFS to be calculated. Therefore, CHFS score values can range from 0 (least limitation) to 90 (most limitation), with improvements in function or reduction of limitation indicated a decreased score value. The mean change from study entry in CHFS scores at each scheduled assessment are summarized.
Time Frame: Baseline and Months 1, 3, 6, and 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Oral Treprostinil Diethanolamine
Number analyzed (Participants) | 109
units on a scale
  Month 1 | -1.1 (9.7)
  Month 3 | -1.2 (8.7)
  Month 6 | -1.0 (9.3)
  Month 12 | -2.8 (9.7)

4. Primary Outcome: Total Ulcer Number- Mean Change From Time of Study Entry for Each Scheduled Visit Assessment
Description: The total ulcer number includes all ulcers designated as "active", "indeterminate", or "new" for a given visit. The mean change in the total number of ulcers present from time of study entry was summarized for each scheduled visit assessment.
Time Frame: Baseline and Months 1, 3, 6, 9, 12, and 18
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: number of ulcers
Arm/Group | Oral Treprostinil Diethanolamine
Number analyzed (Participants) | 111
number of ulcers
  Month 1 | -0.23 (1.36)
  Month 3 | -0.24 (1.99)
  Month 6 | -0.21 (1.21)
  Month 9 | -0.46 (1.57)
  Month 12 | -0.61 (1.20)
  Month 18 | -1.67 (0.58)

5. Primary Outcome: Formation of New Ulcers
Description: The number and percentage of subjects who developed new ulcers during the study were summarized.
Time Frame: 18 months (or last study visit)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Oral Treprostinil Diethanolamine
Number analyzed (Participants) | 115
participants
  No new ulcers | 48
  At least one new ulcer formed | 63
  Indeterminate / missing data | 4

ADVERSE EVENTS:
Time Frame: 48 months
Arm/Group | Oral Treprostinil Diethanolamine
Serious Adverse Events (participants affected / at risk) | 17/115
Other Adverse Events (participants affected / at risk) | 113/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil Diethanolamine (N=115)
Gastroenteritis (Infections and infestations) | 6 (6)
Infected skin ulcer (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (3)
Pancytopenia (Blood and lymphatic system disorders) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2)
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 1 (1)
Pericardial effusion (Cardiac disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 2 (2)
Femoral artery occlusion (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Impaired gastric emptying (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Renal cell carcinoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Oral Treprostinil Diethanolamine (N=115)
Headache (Nervous system disorders) | 74 (99)
Dizziness (Nervous system disorders) | 22 (24)
Migraine (Nervous system disorders) | 8 (12)
Diarrhea (Gastrointestinal disorders) | 52 (77)
Nausea (Gastrointestinal disorders) | 39 (53)
Vomiting (Gastrointestinal disorders) | 15 (20)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 12 (13)
Constipation (Gastrointestinal disorders) | 9 (9)
Abdominal discomfort (Gastrointestinal disorders) | 7 (10)
Abdominal pain upper (Gastrointestinal disorders) | 7 (9)
Dyspepsia (Gastrointestinal disorders) | 7 (7)
Flatulence (Gastrointestinal disorders) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 (39)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 29 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 19 (27)
Myalgia (Musculoskeletal and connective tissue disorders) | 18 (20)
Back pain (Musculoskeletal and connective tissue disorders) | 11 (12)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 9 (9)
Joint swelling (Musculoskeletal and connective tissue disorders) | 6 (6)
Neck pain (Musculoskeletal and connective tissue disorders) | 6 (7)
Infected skin ulcer (Infections and infestations) | 20 (29)
Localised infection (Infections and infestations) | 15 (18)
Nasopharyngitis (Infections and infestations) | 11 (15)
Influenza (Infections and infestations) | 8 (8)
Sinusitis (Infections and infestations) | 7 (7)
Fatigue (General disorders) | 36 (37)
Oedema peripheral (General disorders) | 18 (20)
Pain (General disorders) | 8 (13)
Pyrexia (General disorders) | 6 (7)
Asthenia (General disorders) | 6 (6)
Skin ulcer (Skin and subcutaneous tissue disorders) | 11 (13)
Pruritus (Skin and subcutaneous tissue disorders) | 9 (10)
Rash (Skin and subcutaneous tissue disorders) | 8 (8)
Flushing (Vascular disorders) | 26 (29)
Cough (Respiratory, thoracic and mediastinal disorders) | 11 (11)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 (12)
Insomnia (Psychiatric disorders) | 18 (19)
Decreased appetite (Metabolism and nutrition disorders) | 11 (11)

LIMITATIONS AND CAVEATS:
Interpretation of the change in digital ulcer status was limited by the lack of a control group and the discontinuation of the study prior to subjects completing all scheduled visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the results of this trial must be consistent with the United Therapeutics publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.